CLINICAL TRIAL: NCT05453305
Title: Venopuncture in Pediatric Emergency Department Using Koala's Distraction Method. Randomized Clinical Trial
Brief Title: Venopuncture in Pediatric Emergency Department Using Koala's Distraction Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PI21/218
Record Dates: First submitted 2022-06-14; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-05

CONDITIONS: Nursing Caries; Emergencies; Venous Puncture
Keywords: Venipuncture; pain; anxiety; stress
MeSH Terms: conditions — Emergencies; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: Traditional venipuncture, on the stretcher. (Active Comparator): the companion will place the child on the stretcher in the supine position with the limb to be punctured in decline. At all times, during the technique, the companion will be present, being able to participate by establishing links of consolation or distraction, as is usually done in the hospital. Simultaneously, a professional from the service will be in charge of holding the chosen extremity, as well as the opposite one. The responsible nurse will perform the venipuncture while another colleague will help with tasks of holding and/or collecting samples.
  Interventions: Procedure: Control group: Traditional venipuncture, on the stretcher.
- Experimental group: DAK method venipuncture, simulating a hug. (Experimental): the caregiver will sit in a chair placing the child on top in front of him, with one leg on each side and the arms resting on the shoulders of the companion. The patient's head will rest on the adult's shoulder, contralateral to the limb to be punctured. Simultaneously, the responsible adult patient will hold the simulating a hug. A professional will take care of immobilizing the chosen limb. The responsible nurse performed the venipuncture while another colleague helped with the tasks of holding and/or collecting samples.
  Interventions: Procedure: Intervention group: DAK method venipuncture, simulating a hug

INTERVENTIONS:
Procedure: Control group: Traditional venipuncture, on the stretcher. — The companion will be given the State/Trait Anxiety Questionnaire(STAI) for the initial assessment of the companion's anxiety and will be asked to recall their perceived emotions during the venipuncture. The observer will assess child pain and stress using FLACC and Groningen scale and will record it. Next, the companion will place the child on the stretcher in supine position with the limb to be punctured in decline. During the technique, the companion will be present, being able to participate by establishing links of consolation or distraction, as is usually done in the hospital. Simultaneously, a professional from the service will be in charge of holding the chosen extremity, as well as the opposite one. The responsible nurse will perform the venipuncture and/or collecting samples. The observer will assess child's pain and stress and caregiver's STAI during the intervention with the same scales.
  Arms: Control group: Traditional venipuncture, on the stretcher.
Procedure: Intervention group: DAK method venipuncture, simulating a hug — The companion will be given the State/Trait Anxiety Questionnaire(STAI) for the initial evaluation of the companion's anxiety and will be asked to recall their perceived emotions during the venipuncture. The observer will assess child's pain and stress using the FLACC and Groningen scale and record it. Subsequently, the caregiver will sit in a chair placing the child on top in front of him, with one leg on each side and the arms resting on the shoulders of the companion. The patient's head will rest on the adult's shoulder, contralateral to the limb to be punctured. Simultaneously, the responsible adult patient will hold the simulating a hug. A professional will take care of immobilizing the chosen limb. The responsible nurse performed the venipuncture and collecting samples. The observer will assess the child's pain and stress during the intervention, and will deliver the STAI to the caregiver, to be completed with their perceived sensations during the technique.
  Arms: Experimental group: DAK method venipuncture, simulating a hug.

SUMMARY:
A randomized clinical trial will be performed. Patients aged 3 and 4 years who attend the pediatric emergency service of the Miguel Servet Hospital in Zaragoza and require venipuncture will be selected. In the control group, traditional venipuncture will be performed, placing the child in supine position on the stretcher with the limb to be punctured in decline. In the intervention group, the DAK method will be used, where the adult will hold the child simulating a hug. A professional will take care of immobilizing the chosen limb, and the nurse will perform the venipuncture. The researchers believe that 3 and 4-year-old children subjected to venipuncture using the Koala Attachment Distraction method present a lower level of stress and pain, as well as their companions a lower level of anxiety, compared to those subjected to physical restraint.

Condition of disease: Patients aged 3 and 4 years, who attend the pediatric emergency service of the Miguel Servet Hospital in Zaragoza and require venipuncture.

Intervention: Traditional venipuncture, in supine position on the stretcher with the limb to be punctured in decline. + DAK method, simulating a hug.

DETAILED DESCRIPTION:
A randomized clinical trial will be performed. 220 participants between 3 and 4 years old will be selected and randomized to participate. Control group and experimental group will enrolled 110 participants each one. Control group will be venipunctured in the traditional way. Intervention group will be venipunctured using the DAK method. Before and during the venipuncture, three tests will be performed. To assess level's pain, before and during the technique, the Face, Legs, Activity and Consolability (FLACC) scale will be used, obtaining an assessment of maximum, severe, moderate, mild or no pain.

To evaluate the child's stress, before and during the technique, the Groningen Anxiety Scale will be used, which assesses 3 items: the child's condition, muscle tension and crying, classifying them in 5 degrees from least to greatest stress. To assess the perceived anxiety of the companion, the State-Trait Anxiety Inventory (STAI) questionnaire will be used, classifying it in percentiles according to age and sex. In both groups, a trained observer will evaluate the child's pain and stress before and during the technique, and the companion will fill out the STAI questionnaire. Study participants will be required to read an information sheet and sign an informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 and 4 years who require venipuncture in the Emergency Department.
* To signature of the informed consent by the patient's companion.

Exclusion Criteria:

* Children with psychomotor retardation, due to difficulties in assessing stress and pain in this group of patients.
* Cancer patients with subcutaneous reservoir.
* Patients with diabetes mellitus or other pathologies that imply alterations in the sensitivity of the skin.
* Children classified as priority level I or II in triage.
* Children with special needs and/or classified as "minimum waiting".
* Children with an inability to understand and express the language (linguistic barrier).
* Previous administration of analgesic, sedative or relaxing drugs.
* Prior venipuncture less than 24 hours.

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
To measure changes in the child's pain during venipuncture using the Koala Attachment Distraction (DAK) method. | Two time points: Baseline (previous venipuncture) and during procedure (blood draw)
  The observer will assess child pain using Face, Legs, Activity and Consolability (FLACC) scale, each category is scored 0-2. Total score goes from 0, which indicates relaxed and comfortable to 10, severe pain.
To measure changes in the child's stress during venipuncture using the Koala Attachment Distraction (DAK) method. | Two time points: Baseline (previous venipuncture) and during procedure (blood draw)
  Stress will be recorded with Groningen Distress Scale (GDS) which goes from 1 (calm not cry) to 5 (agitated, physical resistance y screaming).

SECONDARY OUTCOMES:
To measure changes in the level of pain in the child's venipunctured using physical restraint and compare to the DAK method. | Two time points: Baseline (previous venipuncture) and during procedure (blood draw)
  The observer will assess child pain using Face, Legs, Activity and Consolability (FLACC) scale, each category is scored 0-2. Total score goes from 0, which indicates relaxed and comfortable to10, severe pain.
To measure changes in the level of stress in the child's venipunctured using physical restraint and compare to the DAK method. | Two time points: Baseline (previous venipuncture) and during procedure (blood draw)
  Stress will be recorded with Groningen Distress Scale (GDS) which goes from 1 (calm not cry) to 5 (agitated, physical resistance y screaming).
To measure the changes in the level of perceived anxiety of companions when performing venipuncture with the DAK method and physical restraint. | Two time points: Baseline (previous venipuncture) and immediately after procedure (blood draw), where companion must recall their perceived emotions during venipuncture.
  The companion will be given the State part of the State/Trait Anxiety Questionnaire(STAI) Result goes from 0 to 30, being higher scores higher anxiety levels.

CONTACTS AND LOCATIONS:
Overall Officials: Tania Fernández, Nursing, Principal Investigator — Hospital Universitario Miguel Servet (Zaragoza, Spain)
Locations (1):
- Hospital Universitario Miguel Servet, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ali S, McGrath T, Drendel AL. An Evidence-Based Approach to Minimizing Acute Procedural Pain in the Emergency Department and Beyond. Pediatr Emerg Care. 2016 Jan;32(1):36-42; quiz 43-4. doi: 10.1097/PEC.0000000000000669. PMID 26720064
- [Result] Hartling L, Newton AS, Liang Y, Jou H, Hewson K, Klassen TP, Curtis S. Music to reduce pain and distress in the pediatric emergency department: a randomized clinical trial. JAMA Pediatr. 2013 Sep;167(9):826-35. doi: 10.1001/jamapediatrics.2013.200. PMID 23857075
- [Result] Shave K, Ali S, Scott SD, Hartling L. Procedural pain in children: a qualitative study of caregiver experiences and information needs. BMC Pediatr. 2018 Oct 13;18(1):324. doi: 10.1186/s12887-018-1300-y. PMID 30316301
- [Result] Thompson S, Ayers S, Pervilhac C, Mahoney L, Seddon P. The association of children's distress during venepuncture with parent and staff behaviours. J Child Health Care. 2016 Sep;20(3):267-76. doi: 10.1177/1367493515598643. Epub 2015 Aug 27. PMID 26316521
- [Result] Yoo H, Kim S, Hur HK, Kim HS. The effects of an animation distraction intervention on pain response of preschool children during venipuncture. Appl Nurs Res. 2011 May;24(2):94-100. doi: 10.1016/j.apnr.2009.03.005. Epub 2009 Jul 15. PMID 20974061
- [Result] Bailey B, Trottier ED. Managing Pediatric Pain in the Emergency Department. Paediatr Drugs. 2016 Aug;18(4):287-301. doi: 10.1007/s40272-016-0181-5. PMID 27260499
- [Result] Bahorski JS, Hauber RP, Hanks C, Johnson M, Mundy K, Ranner D, Stoutamire B, Gordon G. Mitigating procedural pain during venipuncture in a pediatric population: A randomized factorial study. Int J Nurs Stud. 2015 Oct;52(10):1553-64. doi: 10.1016/j.ijnurstu.2015.05.014. Epub 2015 Jun 10. PMID 26118441
- [Result] Garcia-Aracil N, Ramos-Pichardo JD, Castejon-de la Encina ME, Jose-Alcaide L, Julia-Sanchis R, Sanjuan-Quiles A. Effectiveness of non-pharmacological measures for reducing pain and fear in children during venipuncture in the emergency department: a vibrating cold devices versus distraction. Emergencias. 2018 Jun;30(3):182-185. English, Spanish. PMID 29687673
- [Result] Vagnoli L, Caprilli S, Vernucci C, Zagni S, Mugnai F, Messeri A. Can presence of a dog reduce pain and distress in children during venipuncture? Pain Manag Nurs. 2015 Apr;16(2):89-95. doi: 10.1016/j.pmn.2014.04.004. Epub 2014 Nov 4. PMID 25439114
- [Result] Canbulat N, Ayhan F, Inal S. Effectiveness of external cold and vibration for procedural pain relief during peripheral intravenous cannulation in pediatric patients. Pain Manag Nurs. 2015 Feb;16(1):33-9. doi: 10.1016/j.pmn.2014.03.003. Epub 2014 Jun 7. PMID 24912740
- [Result] Brenner SM, Rupp V, Boucher J, Weaver K, Dusza SW, Bokovoy J. A randomized, controlled trial to evaluate topical anesthetic for 15 minutes before venipuncture in pediatrics. Am J Emerg Med. 2013 Jan;31(1):20-5. doi: 10.1016/j.ajem.2012.05.003. Epub 2012 Jul 16. PMID 22809774
- [Result] Oliveira NC, Santos JL, Linhares MB. Audiovisual distraction for pain relief in paediatric inpatients: A crossover study. Eur J Pain. 2017 Jan;21(1):178-187. doi: 10.1002/ejp.915. Epub 2016 Jul 26. PMID 27461092
- [Result] Pillai Riddell RR, Racine NM, Turcotte K, Uman LS, Horton RE, Din Osmun L, Ahola Kohut S, Hillgrove Stuart J, Stevens B, Gerwitz-Stern A. Non-pharmacological management of infant and young child procedural pain. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD006275. doi: 10.1002/14651858.CD006275.pub2. PMID 21975752